CLINICAL TRIAL: NCT01430091
Title: Relative Bioavailability of a Prasugrel Paediatric Orally Disintegrating Tablet Formulation Compared to the Tablet in Healthy Adult Subjects
Brief Title: A Relative Bioavailability Study of a Prasugrel Orally Disintegrating Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13040; H7T-EW-TADQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-09-06; First posted 2011-09-07 (Estimated); Results first posted 2012-11-06 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-10

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Prasugrel clinical formulation (Active Comparator): A single 5-milligram (mg) prasugrel tablet administered orally by swallowing it whole on 1 occasion.
  Interventions: Drug: Prasugrel (clinical formulation)
- Prasugrel (ODT) - on tongue (Experimental): A single 5-mg prasugrel orally disintegrating tablet (ODT) administered orally by placing it on top of the tongue and keeping it there until it disintegrates.
  Interventions: Drug: Prasugrel (Orally Disintegrating Tablet [ODT])
- Prasugrel (ODT) - apple juice (Experimental): A single 5-mg prasugrel ODT administered orally by placing it on top of the tongue followed by drinking approximately 180 milliliters (ml) apple juice within 1 minute after the tablet finishes disintegration.
  Interventions: Drug: Prasugrel (Orally Disintegrating Tablet [ODT])
- Prasugrel (ODT) - chewed (Experimental): A single 5-mg prasugrel ODT administered orally by placing it on top of the tongue, but then chewed and swallowed rather than waiting for it to disintegrate.
  Interventions: Drug: Prasugrel (Orally Disintegrating Tablet [ODT])
- Prasugrel (ODT) - under tongue (Experimental): A single 5-mg prasugrel ODT administered orally by placing it under (rather than on top of) the tongue and keeping it there until it disintegrates.
  Interventions: Drug: Prasugrel (Orally Disintegrating Tablet [ODT])

INTERVENTIONS:
Drug: Prasugrel (clinical formulation) — Administered orally
  Other Names: LY640315; Effient®; Efient®
  Arms: Prasugrel clinical formulation
Drug: Prasugrel (Orally Disintegrating Tablet [ODT]) — Administered orally
  Other Names: LY640315; Effient®; Efient®
  Arms: Prasugrel (ODT) - apple juice; Prasugrel (ODT) - chewed; Prasugrel (ODT) - on tongue; Prasugrel (ODT) - under tongue

SUMMARY:
This study compares the clinical tablet formulation of prasugrel taken orally with an orally disintegrating tablet (ODT) taken orally. The study will evaluate the amount of prasugrel active metabolite circulating in the blood for each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females, as determined by medical history and physical examination
* Are either women who are of child-bearing potential, surgically sterilised or defined as post-menopausal. Female subjects of child-bearing potential (not surgically sterilised between menarche and menopause) must have a negative pregnancy test at the time of screening and must be using a reliable method of birth control. These include tubal ligation, an intrauterine device which has been in place for at least 3 months, the oral contraceptive pill which has been taken, without difficulty, for at least 3 months, or an approved hormonal implant. Barrier methods alone (condoms or diaphragm/cap) are not acceptable, but must be used in conjunction with a chemical method, that is, spermicidal gel. A woman is presumed to be post-menopausal if she has had amenorrhoea for greater than 12 months alone or amenorrheic for 6 to 12 months and has a serum oestradiol concentration <73 picomoles per liter (pmol/L) (20 picograms per milliliter [pg/mL]) (not applicable for women on hormone replacement therapy [HRT; oestrogen]) and a follicle stimulating hormone (FSH) concentration >40 international units per liter (IU/L).
* Have clinical laboratory test results within normal reference range for the investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Between the body mass index (BMI) of 18.5 and 32.0 kilograms per meter squared (kg/m^2), inclusive
* Have acceptable blood pressure (BP) and heart rate (HR) (supine) as determined by the investigator
* Have venous access sufficient to allow blood sampling
* Are reliable and willing to make themselves available for the duration of the study, and will abide by the research unit policy and procedure and study restrictions
* Have given written informed consent approved by Lilly and the Ethical Review Board (ERB) governing the site

Exclusion Criteria:

* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, haematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data, as determined by the investigator
* Evidence of significant active neuropsychiatric disease
* Have a history or presence of significant bleeding disorders, that is, haematemesis, melaena, severe or recurrent epistaxis, haemoptysis, haemorrhage, clinically overt haematuria, or intracranial haemorrhage
* Have a history (within the last 5 years) or presence of gastric ulcers. Previous history of duodenal ulcer is acceptable but must have been successfully surgically or medically treated with no further evidence of disease in the past 6 months (from screening)
* Have a personal or family history of coagulation or bleeding disorders or reasonable suspicion of vascular malformations, for example, cerebral haemorrhage, aneurysm, or premature stroke (cerebrovascular accident <65 years of age)
* Have a self-reported history of significant bleeding from trauma (for example, prolonged bleeding after tooth extraction)
* Are pre-menopausal females with a history or presence of menorrhagia within the last 5 years (from screening)
* Have clinically significant out of range values for prothrombin time (PT), activated partial thromboplastin time (APTT), or platelet count at screening
* Have repeatedly reported positive results (at least 2 separate samples) on the faecal occult blood examination
* Have a history of major surgery within 3 months of screening
* Have planned surgery within 14 days after the last study day
* Have a clinically significant abnormality in fundoscopic examination or petechiae examination
* Have any other clinically significant abnormality following the investigator's review of the prestudy physical examination, electrocardiogram (ECG) and clinical (safety) laboratory tests
* Regularly use known drugs of abuse and/or show unacceptable positive findings on urinary drug screening
* Have known allergies or significant hypersensitivity to prasugrel or related drugs, or a history of relevant allergic drug reactions of any origin
* Have donated blood of more than 500 mL within the previous 1 month before prasugrel administration
* Show evidence of positive human immunodeficiency virus (HIV) antibodies
* Show evidence of positive hepatitis C antibody
* Show evidence of positive hepatitis B surface antigen
* Have a regular alcohol intake greater than 21 units/week for males or 14 units/week for females or are unwilling to comply with the alcohol consumption requirements from 48 hours prior to the first dose of prasugrel until discharge from the clinical research unit (CRU) after the final Pharmacokinetics (PK) sample of Period 5 has been taken. One unit of alcohol is equal to 8 g ethanol
* Smoke 10 or more cigarettes per day
* Use prescription, over the counter or herbal medications that cannot safely be discontinued within 14 days prior to prasugrel administration. Exceptions: subjects may continue thyroid replacement therapy, HRT (oestrogen), contraceptives and certain medications that are inhaled or applied to the skin, eyes, or nose. The influenza vaccine may also be administered; however this must be at least 72 hours before any prasugrel dose
* Use proton pump inhibitors, antacids, or H2 antagonists, which may impact stomach pH
* Have participated in a study involving administration of an investigational compound within the 30 days prior to prasugrel administration
* Have any other condition that, in the opinion of the principal investigator increases the risk to the study subject or decreases the likelihood of obtaining reliable results from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants: Received 5 milligrams (mg) prasugrel as either the clinical tablet or as an orally disintegrating tablet (ODT).
Period: Overall Study
Arm/Group | Participants
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants: Total Number of Study Participants
Arm/Group | Participants
Number analyzed (Participants) | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 37.1 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 11
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve From Time Zero to the Last Measureable Concentration (AUC[0-tlast]) of Prasugrel's Active Metabolite (PRAS-AM)
Time Frame: Pre-dose up to 8 hours post-dose after each treatment
Population: Pharmacokinetic analyses were conducted on the full analysis set, which included all data from all randomized participants receiving at least 1 dose of prasugrel.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram * hour per milliliter (ng*h/mL)
Groups:
- Clinical Tablet: 5-milligrams (mg) prasugrel clinical tablet swallowed whole with approximately 180 milliliters (ml) water.
- ODT on Top of Tongue: 5-mg prasugrel orally disintegrating tablet (ODT) placed on the tongue and allowed to disintegrate, no liquid given.
- ODT on Top of Tongue With Juice Chaser: 5-mg prasugrel ODT placed on the tongue and allowed to disintegrate, followed by approximately 180 milliliters (ml) apple juice chaser.
- ODT Chewed and Swallowed: 5-mg prasugrel ODT chewed and swallowed, no liquid given.
- ODT Placed Under the Tongue: 5-mg prasugrel ODT placed under the tongue and allowed to disintegrate, no liquid given.
Arm/Group | Clinical Tablet | ODT on Top of Tongue | ODT on Top of Tongue With Juice Chaser | ODT Chewed and Swallowed | ODT Placed Under the Tongue
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18
nanogram * hour per milliliter (ng*h/mL) | 43.3 (27.0) | 42.7 (25.0) | 42.3 (29) | 41.0 (32) | 42.0 (30)

2. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Prasugrel's Active Metabolite (PRAS-AM)
Time Frame: Pre-dose up to 8 hours post-dose after each treatment
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Clinical Tablet | ODT on Top of Tongue | ODT on Top of Tongue With Juice Chaser | ODT Chewed and Swallowed | ODT Placed Under the Tongue
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18
nanogram per milliliter (ng/mL) | 47.3 (48) | 47.6 (19) | 32.3 (37) | 38.3 (47) | 41.9 (37)

3. Primary Outcome: Pharmacokinetics: Time of Maximum Concentration (Tmax) of Prasugrel's Active Metabolite (PRAS-AM)
Time Frame: Pre-dose up to 8 hours post-dose after each treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Groups:
- Clinical Tablet: 5-milligrams (mg) prasugrel clinical tablet swallowed whole approximately 180 milliliters (ml) with water.
- ODT on Top of Tongue: 5-mg prasugrel orally disintegrating table (ODT) placed on the tongue and allowed to disintegrate, no liquid given.
Arm/Group | Clinical Tablet | ODT on Top of Tongue | ODT on Top of Tongue With Juice Chaser | ODT Chewed and Swallowed | ODT Placed Under the Tongue
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18
hours | 0.50 [0.25 to 1.00] | 0.50 [0.25 to 2.00] | 0.75 [0.25 to 1.50] | 0.75 [0.25 to 2.00] | 0.50 [0.25 to 2.00]

ADVERSE EVENTS:
Groups:
- ODT (Top of Tongue): 5-mg prasugrel orally disintegrating tablet (ODT) placed on the tongue and allowed to disintegrate, no liquid given.
- ODT (Juice Chaser): 5-mg prasugrel ODT placed on the tongue and allowed to disintegrate, followed by approximately 180 milliliters (ml) apple juice chaser.
- ODT (Chew and Swallow): 5-mg prasugrel ODT chewed and swallowed, no liquid given.
- ODT (Under Tongue): 5-mg prasugrel ODT placed under the tongue and allowed to disintegrate, no liquid given.
Arm/Group | Clinical Tablet | ODT (Top of Tongue) | ODT (Juice Chaser) | ODT (Chew and Swallow) | ODT (Under Tongue)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/18 | 3/18 | 1/18 | 0/18 | 0/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical Tablet (N=18) | ODT (Top of Tongue) (N=18) | ODT (Juice Chaser) (N=18) | ODT (Chew and Swallow) (N=18) | ODT (Under Tongue) (N=18)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days